CLINICAL TRIAL: NCT04286386
Title: Development &Amp; Evaluation of a Quantitative HP MRI Clinical Prostate Cancer Exam
Brief Title: Development and Evaluation of a Quantitative HP MRI for Clinical Prostate Cancer Exam
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-1164; NCI-2020-00746 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-1164 (Other: M D Anderson Cancer Center); R01CA211150 (NIH)
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Prostate Adenocarcinoma
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm Ia (MRSI): Patients receive hyperpolarized carbon C 13 pyruvate IV and undergo MRSI at least 5 weeks after prostate cancer biopsy.
  Interventions: Other: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Spectroscopic Imaging
- Arm Ib (MRSI): Patients receive hyperpolarized carbon C 13 pyruvate IV and undergo MRSI at least 5 weeks after prostate cancer biopsy and at a second time 3-4 weeks after.
  Interventions: Other: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Spectroscopic Imaging
- Arm II (MRSI, surgery): Patients receive hyperpolarized carbon C 13 pyruvate IV and undergo MRSI at least 5 weeks after prostate cancer biopsy, followed by standard of care surgery within 6 months after.
  Interventions: Other: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Spectroscopic Imaging; Procedure: Surgical Procedure

INTERVENTIONS:
Other: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized 13C-Pyruvate; Hyperpolarized Pyruvate (13C)
Procedure: Magnetic Resonance Spectroscopic Imaging — Undergo MRSI
  Other Names: 1H- Nuclear Magnetic Resonance Spectroscopic Imaging; 1H-nuclear magnetic resonance spectroscopic imaging; Magnetic Resonance Spectroscopy; MRS; MRS Imaging; MRSI; proton magnetic resonance spectroscopic imaging
Procedure: Surgical Procedure — Undergo standard of care surgery
  Other Names: Operation; surgery; Surgical; Surgical Interventions; Surgical Procedures; Type of Surgery
  Groups: Arm II (MRSI, surgery)

SUMMARY:
This trial examines if a prostate magnetic resonance spectroscopic imaging can be performed on a 3T scanner using an investigational contrast called hyperpolarized 13-C pyruvate for the development of a clinical prostate cancer exam. 3T refers to the strength of the magnetic resonance spectroscopic imaging (MRSI) machine. MRSI is a magnetic resonance imaging (MRI) technique that can show certain chemical differences in healthy and diseased prostate tumor tissue compared to standard multiparametric MRI that may not detect the tumor. Hyperpolarized (HP) 13-C pyruvate is a contrast drug that may help the scanner see the tumor site better during imaging. Hyperpolarization of 13-C pyruvate may allow pyruvate and its metabolites to be detected upon injection, which in turn, allow the prostate cancer to be found and treated.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess reproducibility of quantitative spectroscopic and imaging parameters in hyperpolarized 13-C pyruvate magnetic resonance spectroscopic imaging (MRSI), including kpl, which assesses the rate of conversion of 13-C pyruvate to 13-C lactate in the tissue of interest, using a test-retest study design.

II. To test the reproducibility of the normalized area under the lactate curve (nLac), a semi-quantitative biomarker for tumor metabolism.

SECONDARY OBJECTIVES:

I. To provide initial assessment of the sensitivity and specificity of hyperpolarized 13-C-pyruvate MRSI performed pre-therapy for detecting high risk localized prostate cancer.

II. To assess the correlation between kpl and tumor grade.

OUTLINE: Patients are assigned to 1 of 3 arms.

ARM Ia: Patients receive hyperpolarized carbon C 13 pyruvate intravenously (IV) and undergo MRSI at least 5 weeks after prostate cancer biopsy.

ARM Ib: Patients receive hyperpolarized carbon C 13 pyruvate IV and undergo MRSI at least 5 weeks after prostate cancer biopsy and at a second time 3-4 weeks after.

ARM II: Patients receive hyperpolarized carbon C 13 pyruvate IV and undergo MRSI at least 5 weeks after prostate cancer biopsy, followed by standard of care surgery within 6 months after.

After the completion of study, patients in Arm Ia and Arm Ib are followed up once.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate adenocarcinoma (Arm 1 & 2)
* Clinically appropriate for active surveillance (Arm 1)
* Prior prostate biopsy must have been performed at least 5 weeks prior imaging (Arm 1 & 2)
* Patient must be scheduled to undergo radical prostatectomy within 6 months of multi-parametric magnetic resonance imaging (MP-MRI) + hyperpolarized (HP) [1-13C]-pyruvate imaging, consistent with American College of Radiology Imaging Network (ACRIN) Protocol: ACRIN 6659 (Arm 2)
* At least 10% of enrolled patients will have high risk of disease progression (Cancer of the Prostate Risk Assessment - [CAPRA] 6-10) and no more than 50% of enrolled patients will have low risk of progression (CAPRA < 3) (Arm 2)

Exclusion Criteria:

* Contraindication to MRI (Arm 1 & 2)
* Allergy to gadavist intravenous contrast (Arm 1 & 2)
* Any known medical history of arrhythmias such as atrial fib, etc. (Arm 1 & 2)
* Prior therapy for prostate cancer, except for 5-alpha reductase inhibitor discontinued at least one month prior to imaging (Arm 1 & 2)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven prostate cancer that are enrolled in an active surveillance protocol, and patients that are scheduled for prostatectomy at MD Anderson
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of the kpl measurement | 3 years
  Will be assessed using a test-retest study design. Will be summarized by the intra-class correlation coefficient (ICC). Data from patients at both MD Anderson and University of San Fransisco, San Fransisco (UCSF) will be pooled if possible to increase significance. Bland-Altman analysis will be included if the ICC proves unreliable as a measure of reproducibility. ICC is sensitive to data range; thus, Bland-Altman plot, limits of agreement, repeatability coefficient, and the within-patient coefficient of variation (wCV) may be included as appropriate.
Reproducibility of the normalized area under the lactate curve (nLac) | 3 years
  Will be carried out using data from N=40 patients on active surveillance at MD Anderson. Will be summarized by the ICC. Data from patients at both MD Anderson and University of San Fransisco, San Fransisco (UCSF) will be pooled if possible to increase significance. Bland-Altman analysis will be included if the ICC proves unreliable as a measure of reproducibility. ICC is sensitive to data range; thus, Bland-Altman plot, limits of agreement, repeatability coefficient, and the within-patient coefficient of variation (wCV) may be included as appropriate.

SECONDARY OUTCOMES:
Specificity of HP 13-C-pyruvate MRSI for detecting high risk localized prostate cancer | 3 years
  Analysis will be restricted to lesions > 0.5 cc and the 3 most significant pathologic cancer foci from each patient. Specificity will be calculated as the ratio of true negatives to the sum of true negatives and false positives. Specificity will be assessed using pooled data from MD Anderson (N=25) and UCSF (N=25). A ROC analysis will be carried out.
Sensitivity of hyperpolarized (HP) 13-C-pyruvate magnetic resonance spectroscopy imaging (MRSI) for detecting high risk localized prostate cancer | 3 years
  Analysis will be restricted to lesions > 0.5 cc and the 3 most significant pathologic cancer foci from each patient. Sensitivity will be calculated as the ratio of true positives (matches) to the sum of true positives and false negatives. Sensitivity will be assessed using pooled data from MD Anderson (N=25) and UCSF (N=25). A receiver operating characteristic (ROC) analysis will be carried out.
Kpl | 3 years
  Correspondence between kpl, imaging biomarkers from the multiparametric MRI exam, and tumor grade will be assessed. Imaging biomarkers will be compared with pathologic grade (benign, Epstein grade grouping 1; intermediate, Epstein 2-3; and high-grade, Epstein 4-5) using analysis of variance (ANOVA) with Newman-Keuls post-hoc test to determine associations.

CONTACTS AND LOCATIONS:
Overall Officials: Tharakeswara Bathala, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org